CLINICAL TRIAL: NCT02692755
Title: Phase II Safety Study of Palbociclib in Combination With Letrozole or Fulvestrant in African American Women With Hormone Receptor Positive HER2 Negative Advanced Breast Cancer
Brief Title: Palbociclib / Letrozole or Fulvestrant in African American Women With HR+ HER2- Breast Cancer
Acronym: PALINA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: University of Chicago (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1396
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Results first posted 2021-08-20 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-08

CONDITIONS: Hormone Receptor Positive HER-2 Negative Breast Cancer
Keywords: African American
MeSH Terms: interventions — palbociclib; Letrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palbociclib + Letrozole or Fulvestrant (Experimental)
  Interventions: Drug: Palbociclib + Letrozole or Fulvestrant

INTERVENTIONS:
Drug: Palbociclib + Letrozole or Fulvestrant — Palbociclib x 21 days with a 7 day rest plus 2.5 mg Letrozole QD (no break) or Fulvestrant 500mg IM every 2 weeks for 3 doses and then every 4 weeks until progression or maximum of 12 months
  Other Names: Ibrance; Femara; Faslodex

SUMMARY:
This study aims to evaluate the hematological safety of palbociclib with letrozole and fulvestrant in African American women with hormone receptor positive HER2 negative advanced breast cancer. Hematological safety is a composite endpoint of episodes of febrile neutropenia and treatment discontinuation due to neutropenia according to current recommendations for management of neutropenia

DETAILED DESCRIPTION:
The study is designed to assess the rate of completion of planned oncology therapy in the absence of a hematological event defined as episodes of febrile neutropenia and treatment discontinuation due to neutropenia. A completion rate of 80% is considered of clinical relevance as to benefit breast cancer patients who are at a higher risk of having ethnic neutropenia where as a completion rate of 60% is considered poor and to justify additional safety studies. A two stage design with a total of 35 patients is used to test if the completion rate is at least 80% versus if it is below 60% with 80% power at a significance level of 5%.

An exact confidence interval of the completion rate will be calculated. Investigators estimate there will be no more than a 10% rate of febrile neutropenia. Due to the small sample size, the analysis of secondary endpoints will be descriptive and will not include specific hypothesis testing.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identified Black, African or African American women of ≥ 18 years of age with proven diagnosis of advanced adenocarcinoma of the breast (locoregionally recurrent or metastatic disease)
2. ER-positive and/or PgR-positive tumor based on local laboratory results
3. HER2-negative breast cancer based on local laboratory results (test to be used as per local practice)
4. Patients must be appropriate candidates for letrozole or fulvestrant therapy
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
6. Adequate bone marrow function:

   * Absolute Neutrophil Count (ANC) ≥ 1,000/mm3 (1.0 x 109/L);
   * Platelets ≥100,000/mm3 (100 x 109/L);
   * Hemoglobin ≥9 g/dL (90 g/L).

Exclusion Criteria:

1. Current use of food or drugs known to be potent inhibitors or inducers of CYP3A4
2. Active uncontrolled or symptomatic brain metastases. Previously treated and clinically stable, as per Investigator's judgment, brain metastases are permitted.
3. Previous CDK4/6 inhibitor

   -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2021-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Isaacs, MD, Principal Investigator — MedStar Georgetown University Hospital
Locations (6):
- United States (6):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of chemotherapy and hormonal therapy for early breast cancer on recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 May 14-20;365(9472):1687-717. doi: 10.1016/S0140-6736(05)66544-0. PMID 15894097
- [Background] Wood WC, Muss HB, Solin LJ, Olopade OI. Malignant Tumors of the Breast. In: DeVita VT Jr, Hellmann S, Rosenberg SA, editors. Cancer, Principle and Practice of Oncology, 7thEdition, Lippincott Williams and Wilkins; 2005; 1415-1477.
- [Background] Leung BS, Potter AH. Mode of estrogen action on cell proliferation in CAMA-1 cells: II. Sensitivity of G1 phase population. J Cell Biochem. 1987 Jul;34(3):213-25. doi: 10.1002/jcb.240340307. PMID 3611201
- [Background] Sutherland RL, Hall RE, Taylor IW. Cell proliferation kinetics of MCF-7 human mammary carcinoma cells in culture and effects of tamoxifen on exponentially growing and plateau-phase cells. Cancer Res. 1983 Sep;43(9):3998-4006. PMID 6871841
- [Background] Mouridsen H, Gershanovich M, Sun Y, Perez-Carrion R, Boni C, Monnier A, Apffelstaedt J, Smith R, Sleeboom HP, Jaenicke F, Pluzanska A, Dank M, Becquart D, Bapsy PP, Salminen E, Snyder R, Chaudri-Ross H, Lang R, Wyld P, Bhatnagar A. Phase III study of letrozole versus tamoxifen as first-line therapy of advanced breast cancer in postmenopausal women: analysis of survival and update of efficacy from the International Letrozole Breast Cancer Group. J Clin Oncol. 2003 Jun 1;21(11):2101-9. doi: 10.1200/JCO.2003.04.194. PMID 12775735
- [Background] Finn RS, Dering J, Conklin D, Kalous O, Cohen DJ, Desai AJ, Ginther C, Atefi M, Chen I, Fowst C, Los G, Slamon DJ. PD 0332991, a selective cyclin D kinase 4/6 inhibitor, preferentially inhibits proliferation of luminal estrogen receptor-positive human breast cancer cell lines in vitro. Breast Cancer Res. 2009;11(5):R77. doi: 10.1186/bcr2419. PMID 19874578
- [Background] Schwartz GK, LoRusso PM, Dickson MA, Randolph SS, Shaik MN, Wilner KD, Courtney R, O'Dwyer PJ. Phase I study of PD 0332991, a cyclin-dependent kinase inhibitor, administered in 3-week cycles (Schedule 2/1). Br J Cancer. 2011 Jun 7;104(12):1862-8. doi: 10.1038/bjc.2011.177. Epub 2011 May 24. PMID 21610706
- [Background] Flaherty KT, Lorusso PM, Demichele A, Abramson VG, Courtney R, Randolph SS, Shaik MN, Wilner KD, O'Dwyer PJ, Schwartz GK. Phase I, dose-escalation trial of the oral cyclin-dependent kinase 4/6 inhibitor PD 0332991, administered using a 21-day schedule in patients with advanced cancer. Clin Cancer Res. 2012 Jan 15;18(2):568-76. doi: 10.1158/1078-0432.CCR-11-0509. Epub 2011 Nov 16. PMID 22090362
- [Background] DeMichele A, Clark AS, Tan KS, Heitjan DF, Gramlich K, Gallagher M, Lal P, Feldman M, Zhang P, Colameco C, Lewis D, Langer M, Goodman N, Domchek S, Gogineni K, Rosen M, Fox K, O'Dwyer P. CDK 4/6 inhibitor palbociclib (PD0332991) in Rb+ advanced breast cancer: phase II activity, safety, and predictive biomarker assessment. Clin Cancer Res. 2015 Mar 1;21(5):995-1001. doi: 10.1158/1078-0432.CCR-14-2258. Epub 2014 Dec 11. PMID 25501126
- [Background] Finn RS, Crown JP, Lang I, Boer K, Bondarenko IM, Kulyk SO, Ettl J, Patel R, Pinter T, Schmidt M, Shparyk Y, Thummala AR, Voytko NL, Fowst C, Huang X, Kim ST, Randolph S, Slamon DJ. The cyclin-dependent kinase 4/6 inhibitor palbociclib in combination with letrozole versus letrozole alone as first-line treatment of oestrogen receptor-positive, HER2-negative, advanced breast cancer (PALOMA-1/TRIO-18): a randomised phase 2 study. Lancet Oncol. 2015 Jan;16(1):25-35. doi: 10.1016/S1470-2045(14)71159-3. Epub 2014 Dec 16. PMID 25524798
- [Background] A study of Palbociclib (PD-0332991) + letrozole vs. letrozole for first line treatment of postmenopausal women with ER/HER2- advanced breast cancer (PALOMA-2). Available at: https://clinicaltrials.gov/ct2/show/NCT01740427. Accessed on August 9, 2015
- [Background] Turner NC, Huang Bartlett C, Cristofanilli M. Palbociclib in Hormone-Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2015 Oct 22;373(17):1672-3. doi: 10.1056/NEJMc1510345. No abstract available. PMID 26488700
- [Background] NIH Policy and Guidelines on The Inclusion of Women and Minorities as Subjects in Clinical Research - Amended, October, 2001
- [Background] Chen MS Jr, Lara PN, Dang JH, Paterniti DA, Kelly K. Twenty years post-NIH Revitalization Act: enhancing minority participation in clinical trials (EMPaCT): laying the groundwork for improving minority clinical trial accrual: renewing the case for enhancing minority participation in cancer clinical trials. Cancer. 2014 Apr 1;120 Suppl 7(0 7):1091-6. doi: 10.1002/cncr.28575. PMID 24643646
- [Background] Hsieh MM, Everhart JE, Byrd-Holt DD, Tisdale JF, Rodgers GP. Prevalence of neutropenia in the U.S. population: age, sex, smoking status, and ethnic differences. Ann Intern Med. 2007 Apr 3;146(7):486-92. doi: 10.7326/0003-4819-146-7-200704030-00004. PMID 17404350
- [Background] Reich D, Nalls MA, Kao WH, Akylbekova EL, Tandon A, Patterson N, Mullikin J, Hsueh WC, Cheng CY, Coresh J, Boerwinkle E, Li M, Waliszewska A, Neubauer J, Li R, Leak TS, Ekunwe L, Files JC, Hardy CL, Zmuda JM, Taylor HA, Ziv E, Harris TB, Wilson JG. Reduced neutrophil count in people of African descent is due to a regulatory variant in the Duffy antigen receptor for chemokines gene. PLoS Genet. 2009 Jan;5(1):e1000360. doi: 10.1371/journal.pgen.1000360. Epub 2009 Jan 30. PMID 19180233
- [Background] Hsieh MM, Tisdale JF, Rodgers GP, Young NS, Trimble EL, Little RF. Neutrophil count in African Americans: lowering the target cutoff to initiate or resume chemotherapy? J Clin Oncol. 2010 Apr 1;28(10):1633-7. doi: 10.1200/JCO.2009.24.3881. Epub 2010 Mar 1. No abstract available. PMID 20194862
- [Background] Hershman D, Weinberg M, Rosner Z, Alexis K, Tiersten A, Grann VR, Troxel A, Neugut AI. Ethnic neutropenia and treatment delay in African American women undergoing chemotherapy for early-stage breast cancer. J Natl Cancer Inst. 2003 Oct 15;95(20):1545-8. doi: 10.1093/jnci/djg073. PMID 14559877
- [Background] Shajahan-Haq AN, Cheema MS, Clarke R. Application of metabolomics in drug resistant breast cancer research. Metabolites. 2015 Feb 16;5(1):100-18. doi: 10.3390/metabo5010100. PMID 25693144
- [Background] Nowicki S, Gottlieb E. Oncometabolites: tailoring our genes. FEBS J. 2015 Aug;282(15):2796-805. doi: 10.1111/febs.13295. Epub 2015 Apr 30. PMID 25864878
- [Background] Gunther UL. Metabolomics Biomarkers for Breast Cancer. Pathobiology. 2015 Sep;82(3-4):153-65. doi: 10.1159/000430844. Epub 2015 Aug 31. PMID 26330356
- [Background] Shajahan-Haq AN, Cook KL, Schwartz-Roberts JL, Eltayeb AE, Demas DM, Warri AM, Facey CO, Hilakivi-Clarke LA, Clarke R. MYC regulates the unfolded protein response and glucose and glutamine uptake in endocrine resistant breast cancer. Mol Cancer. 2014 Oct 23;13:239. doi: 10.1186/1476-4598-13-239. PMID 25339305
- [Background] Asiago VM, Alvarado LZ, Shanaiah N, Gowda GA, Owusu-Sarfo K, Ballas RA, Raftery D. Early detection of recurrent breast cancer using metabolite profiling. Cancer Res. 2010 Nov 1;70(21):8309-18. doi: 10.1158/0008-5472.CAN-10-1319. Epub 2010 Oct 19. PMID 20959483
- [Background] Lowry MC, Gallagher WM, O'Driscoll L. The Role of Exosomes in Breast Cancer. Clin Chem. 2015 Dec;61(12):1457-65. doi: 10.1373/clinchem.2015.240028. Epub 2015 Oct 14. PMID 26467503
- [Background] Yu S, Cao H, Shen B, Feng J. Tumor-derived exosomes in cancer progression and treatment failure. Oncotarget. 2015 Nov 10;6(35):37151-68. doi: 10.18632/oncotarget.6022. PMID 26452221
- [Background] Yu DD, Wu Y, Zhang XH, Lv MM, Chen WX, Chen X, Yang SJ, Shen H, Zhong SL, Tang JH, Zhao JH. Exosomes from adriamycin-resistant breast cancer cells transmit drug resistance partly by delivering miR-222. Tumour Biol. 2016 Mar;37(3):3227-35. doi: 10.1007/s13277-015-4161-0. Epub 2015 Oct 2. PMID 26432333
- [Background] Lv MM, Zhu XY, Chen WX, Zhong SL, Hu Q, Ma TF, Zhang J, Chen L, Tang JH, Zhao JH. Exosomes mediate drug resistance transfer in MCF-7 breast cancer cells and a probable mechanism is delivery of P-glycoprotein. Tumour Biol. 2014 Nov;35(11):10773-9. doi: 10.1007/s13277-014-2377-z. Epub 2014 Jul 31. PMID 25077924
- [Background] Kelly DL, Kreyenbuhl J, Dixon L, Love RC, Medoff D, Conley RR. Clozapine underutilization and discontinuation in African Americans due to leucopenia. Schizophr Bull. 2007 Sep;33(5):1221-4. doi: 10.1093/schbul/sbl068. Epub 2006 Dec 14. PMID 17170061
- [Background] Xiao JF, Varghese RS, Zhou B, Nezami Ranjbar MR, Zhao Y, Tsai TH, Di Poto C, Wang J, Goerlitz D, Luo Y, Cheema AK, Sarhan N, Soliman H, Tadesse MG, Ziada DH, Ressom HW. LC-MS based serum metabolomics for identification of hepatocellular carcinoma biomarkers in Egyptian cohort. J Proteome Res. 2012 Dec 7;11(12):5914-23. doi: 10.1021/pr300673x. Epub 2012 Nov 1. PMID 23078175
- [Derived] Lynce F, Blackburn MJ, Zhuo R, Gallagher C, Hahn OM, Abu-Khalaf M, Mohebtash M, Wu T, Pohlmann PR, Dilawari A, Tiwari SR, Chitalia A, Warren R, Tan M, Shajahan-Haq AN, Isaacs C. Hematologic safety of palbociclib in combination with endocrine therapy in patients with benign ethnic neutropenia and advanced breast cancer. Cancer. 2021 Oct 1;127(19):3622-3630. doi: 10.1002/cncr.33620. Epub 2021 Jun 22. PMID 34157782

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palbociclib + Letrozole or Fulvestrant
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Palbociclib + Letrozole or Fulvestrant
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 35
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35
HR+/HER2- ABC [Count of Participants; unit: Participants] | 35
Baseline absolute neutrophil count ≥1000/mm3 [Count of Participants; unit: Participants] | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Complete Planned Oncologic Therapy Without the Development of a Hematological Event
Description: For study purpose febrile neutropenia will be defined according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0: "ANC less than 1000/mm3 with a single temperature of >38.3 degrees Celsius (101 degrees Fahrenheit) or a sustained temperature of 38 degrees Celsius (100.4 degrees Fahrenheit) for more than one hour."
  Planned oncology therapy is defined as completion of one year of therapy for advanced breast cancer in the absence of disease progression or cessation of study drug due to progressive disease or non-hematological toxicity.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Letrozole or Fulvestrant
Number analyzed (Participants) | 35
Participants | 35

2. Secondary Outcome: Dose Delays in Palbociclib Attributed to Neutropenia
Description: Number of patients who required dose delays in palbociclib attributed to neutropenia.
Time Frame: 12 months
Population: Including all patients who completed ≥1 treatment cycle
Measure: Count of Participants; unit: Participants
Groups:
- Single ARM: Palbociclib + Letrozole or Fulvestrant
  Palbociclib + Letrozole or Fulvestrant: Palbociclib x 21 days with a 7 day rest plus 2.5 mg Letrozole QD (no break) or Fulvestrant 500mg IM every 2 weeks for 3 doses and then every 4 weeks until progression or maximum of 12 months
Arm/Group | Single ARM
Number analyzed (Participants) | 33
Participants | 17

3. Secondary Outcome: Dose Reductions in Palbociclib Therapy Attributed to Neutropenia
Description: Number of patients who required dose reductions in palbociclib therapy
Time Frame: 12 months
Population: Including all patients who completed ≥1 treatment cycle
Measure: Count of Participants; unit: Participants
Arm/Group | Single ARM
Number analyzed (Participants) | 33
Participants | 13

4. Secondary Outcome: Clinical Benefit Rate
Description: Clinical Benefit Rate (CBR), for those with evaluable disease, defined as the percentage of patients who achieved complete response, partial response and stable disease. RECIST 1.1 was used as the standard way to measure response to treatment. The mean (SD) of specific metabolites were calculated at each time point and graphically assess these measures over time with clinical response and hematological toxicity. The mean change in these variables from baseline to each follow-up point was be calculated. Generalized linear model was utilized for the correlative analysis of clinical response and hematologic events.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single ARM
Number analyzed (Participants) | 33
Participants | 23

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Single ARM
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 8/35
Other Adverse Events (participants affected / at risk) | 32/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single ARM (N=35)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Shortness of breath
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Acute airway obstruction
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — COPD
Suicidal ideation (Psychiatric disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single ARM (N=35)
Abdominal Pain (Gastrointestinal disorders) | 6 (8)
Alkaline Phosphate Increased (Investigations) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 12 (20)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Creatinine increased (Investigations) | 2 (7)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 16 (21)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (9)
Flu like symptoms (General disorders) | 3 (3)
Hot flashes (Vascular disorders) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypertension (Vascular disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (5)
Neutrophil count decreased (Investigations) | 17 (51)
Pain (General disorders) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Platelet count decreased (Investigations) | 4 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
White blood cell decreased (Investigations) | 10 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT02692755/Prot_SAP_000.pdf